CLINICAL TRIAL: NCT06693466
Title: Pain Processing and Pain Assessment in Huntington's Disease a Pilot Study
Brief Title: Huntington's Disease and Pain
Acronym: HD-P1
Status: Not yet recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: European Huntington's Disease Network (Network)
Responsible Party: Principal Investigator, Susanne T de Bot, MD, PhD, Principal Investigator, Leiden University Medical Center
Other Study IDs: P24.014
Record Dates: First submitted 2024-11-05; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Huntington Disease; Pain
Keywords: Huntington's disease; Pain; Pain processing; Pain facilitation; Pain inhibition; Pain Assessment in Impaired Cognition (PAIC15)
MeSH Terms: conditions — Huntington Disease; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adult-onset HD stage 1: The adult-onset HD stage 1 group (total function capacity 11-13) include 10 participants.
  The subjects will be undergo three different pain test batteries .
  Interventions: Other: Facial expression block; Other: Conditioned pain modulation block; Other: Pain facilitation block
- Adult-onset HD stage 2-3: The adult-onset HD stage 2-3 group (total function capacity 3-10) include 10 participants.
  The subjects will be undergo three different pain test batteries .
  Interventions: Other: Facial expression block; Other: Conditioned pain modulation block; Other: Pain facilitation block

INTERVENTIONS:
Other: Facial expression block — Data will be collected to assess the facial expression, body movements and vocalization of (non-) painful heat stimuli. The experiment includes individually tailored and randomly administered painful (perceived as moderate pain) and non-painful heat stimuli.
Other: Conditioned pain modulation block — The conditioned pain modulation will be tested according to internationally agreed standards and includes a painful phasic heat (test stimulus) and a painful tonic cold stimulus (conditioning stimulus).
Other: Pain facilitation block — Pain facilitation will be assessed by using painful mechanical pinprick stimuli. The magnitude of pain experienced after a single mechanical pinprick stimulus is compared to that of a train of 10 pinprick stimuli of the same force.

SUMMARY:
The primary objective of this pilot study is to assess the feasibility of three internationally agreed pain test batteries in patients with Huntington Disease. The pain test batteries are developed to collect data about the facial expression of pain, body movements and vocalization of (non-) painful stimuli, and to collect data for testing the pain inhibition and facilitation. The study population will include 20 patients with genetically confirmed, adult-onset HD, in stage 1 (n=10) and stages 2 - 3 of HD (n = 10).

DETAILED DESCRIPTION:
The primary objective of this pilot study is to assess the feasibility of a comprehensive experimental design with three internationally well-known experimental pain protocols in patients with Huntington Disease.

The exploratory objectives are:

* To explore the psychometric properties (inter-, intra-rater and test-retest reliability and measurement error) of the facial expression, body movements and vocalization items of an observational pain scale, the Pain Assessment in Impaired Cognition Scale (PAIC15), in patients with HD.
* To measure the overall facial expression of pain in patients with HD.
* To explore the prevalence and extent of endogenous pain modulation in HD (facilitation, inhibition and the balance between the two).
* To make an initial estimate of the measurement error (i.e. agreement), stated as the systematic and random error of a patients' score that is not attributed to true changes in the construct to be measured, for each endpoint related in current study to pain processing in HD (e.g. facial expression and the endogenous pain modulation outcomes).

Study design: An experimental, observational, cross-sectional study

Study population: The study population will include 20 patients with genetically confirmed, adult-onset HD, in stage 1 (n=10) and stages 2 - 3 of HD (n = 10).

ELIGIBILITY:
Inclusion Criteria:

1. Genetically and clinically confirmed Adult-onset HD patients (≥ 21 years, CAG repeats ≥ 36; DCL of 4).
2. Good general health apart from having HD. Note: Patients with chronic illness (e.g. hypertension) will be eligible if the illness is stable and well-controlled according to the investigator that will not impact the primary objectives of the study.
3. Able to give written informed consent

Exclusion Criteria:

1. Juvenile and Pediatric Huntington's Disease (age at onset <21 years).
2. Patients in the late stage of the disease (UDHRS-TFC score <3).
3. Have medical, psychiatric, or other conditions (other than HD) that, according to the investigator, may compromise the patient's ability to understand the patient information sheet, to give informed consent, to comply with all study requirements, or to perform study assessments.
4. Have a history of (in the past year) or current (ab)use of any drug, alcohol or medication that, in the opinion of the investigator, may seriously interfere with the primary objectives of the study.
5. The presence of a sensorimotor neuropathy or any another disturbance significantly disturbing the somatosensory systems, based on medical history and/or clinical examination, that can interfere with the pain test battery.
6. Women who are pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genetically and clinically confirmed adult-onset HD patients (AoHD) (clinical onset ≥ 21 years, CAG repeats ≥ 36, Diagnostic Confidence Level [DCL] of 4]), in stage 1 (n=10 [named as HD 1]), stage 2 and 3 of HD (n = 10 [named as HD 2]), according to the Shoulson-Fahn system. Total Function Capacity (TFC) of the Unified Huntington Disease Rating Scale (UHDRS) will be used to define the HD groups: UHDRS-TFC score 11-13 (stage 1), 7-10 (stage 2), 3-6 (stage 3), 1-2 (stage 4) and a score of 0 (stage 5).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The feasibility of a comprehensive experimental design including three different experimental pain protocols in patients with Huntington's Disease | Baseline assessment
  A screening tool was developed to determine whether the comprehensive experimental design, with three various experimental pain protocols, is feasible in patients with HD. After each assessment, the screening tool will be scored. Each item of the screening tool represents an important part of the experimental pain protocol. A 'cut-off' score ranging from 60% to 80% was adopted for each item, indicating the minimum score to be met to consider as feasible for that specific part of the experimental pain protocol.
  The comprehension of the instructions, duration and the completion of the study are examples of items which will be evaluated.

OTHER OUTCOMES:
Psychometric properties of the Pain Assessment in Impaired Cognition- 15 | Baseline assessment - 15 minutes
  The intra-, interrater, test-retest reliability and measurement error (i.e. agreement) of the facial expression, body movements and vocalization items of the Pain Assessment in Impaired Cognition - 15 will be assessed.
  The score of the Pain Assessment in Impaired Cognition - 15 ranges from 0 to 45 points. A score of 4 or higher indicate the presence of possible pain.
Overall facial expression of pain in patients with HD | Baseline assessment - 15 minutes
  The facial expression will be assessed with the Pain Assessment in Impaired Cognition Scale.
  The score on the Pain Assessment in Impaired Cognition Scale ranges from 0 to 45 points. A score of 4 or higher indicate the presence of possible pain.
Conditioned pain modulation | Baseline assessment - 15 minutes
  Pain processing in terms of conditioned pain modulation( pain facilitation, inhibition and the balance between two) will be assessed by the (Computerized) Visual Analogue Scale (CoVAS).
  The (Computerized) Visual Analogue Scale is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A subject marks a point of the line that matches the amount of pain he or she feels.
Conditioned pain modulation | Baseline assessment - 15 minutes
  Pain processing in terms of conditioned pain modulation( pain facilitation, inhibition and the balance between two) will be assessed by the numerical rating scale (NRS) in case the Computerized Visual Analogue Scale is not feasible to use.
  The numerical rating scale consists of a series of numbers rating pain intensity, ranging from 0 to 10, with being 0 being "no pain", and 10 "severe pain".
Measurement error Condition Pain Modulation | Area under the curve; with a time frame 0,1,2,3,4,5,6,7,8,9 to 10 seconds.
  An initial estimate of the measurement error (i.e. agreement) will be tested for the outcome of the endogenous pain modulation.
  The (Computerized) Visual Analogue Scale is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A subject marks a point of the line that matches the amount of pain he or she feels.
  An appropriate analysis will conducted such as (weighted kappa), Intraclass correlation coefficient, SEM and/ or Limits of agreement.
Measurement error Condition Pain Modulation | Difference in mean score of the Numerical Rating Scale. Numerical Rating Scale is scored directly after the stimulus. The duration of the exposure is 10seconds.
  An initial estimate of the measurement error (i.e. agreement) will be tested for the outcome of the endogenous pain modulation.
  The numerical rating scale consists of a series of numbers rating pain intensity, ranging from 0 to 10, with being 0 being "no pain", and 10 "severe pain".
  An appropriate analysis will conducted such as (weighted kappa), Intraclass correlation coefficient, SEM and/ or Limits of agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne de Bot, MD Phd, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Aim is to comply with the standards of the Leiden University Medical Center (LUMC) and the contract of the funder of the study: European Huntington Disease Network (EHDN)

REFERENCES:
- [Background] Yarnitsky D, Granot M, Nahman-Averbuch H, Khamaisi M, Granovsky Y. Conditioned pain modulation predicts duloxetine efficacy in painful diabetic neuropathy. Pain. 2012 Jun;153(6):1193-1198. doi: 10.1016/j.pain.2012.02.021. Epub 2012 Apr 3. PMID 22480803
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039
- [Background] Kunz M, Chatelle C, Lautenbacher S, Rainville P. The relation between catastrophizing and facial responsiveness to pain. Pain. 2008 Nov 15;140(1):127-134. doi: 10.1016/j.pain.2008.07.019. Epub 2008 Sep 9. PMID 18783885
- [Background] Kunz M, de Waal MWM, Achterberg WP, Gimenez-Llort L, Lobbezoo F, Sampson EL, van Dalen-Kok AH, Defrin R, Invitto S, Konstantinovic L, Oosterman J, Petrini L, van der Steen JT, Strand LI, de Tommaso M, Zwakhalen S, Husebo BS, Lautenbacher S. The Pain Assessment in Impaired Cognition scale (PAIC15): A multidisciplinary and international approach to develop and test a meta-tool for pain assessment in impaired cognition, especially dementia. Eur J Pain. 2020 Jan;24(1):192-208. doi: 10.1002/ejp.1477. Epub 2019 Oct 13. PMID 31487411
- [Background] de Waal MWM, van Dalen-Kok AH, de Vet HCW, Gimenez-Llort L, Konstantinovic L, de Tommaso M, Fischer T, Lukas A, Kunz M, Lautenbacher S, Lobbezoo F, McGuire BE, van der Steen JT, Achterberg WP. Observational pain assessment in older persons with dementia in four countries: Observer agreement of items and factor structure of the Pain Assessment in Impaired Cognition. Eur J Pain. 2020 Feb;24(2):279-296. doi: 10.1002/ejp.1484. Epub 2019 Oct 22. PMID 31520424